CLINICAL TRIAL: NCT05535920
Title: A Prospective, Randomized, Multi-Center, Open-Label, Cross-Over Study of Lokelma to Control Interdialytic Hyperkalemia Following Augmentation of Dialysate Potassium
Brief Title: A Prospective, Randomized, Open-Label, Cross-Over Study of Lokelma to Control Interdialytic Hyperkalemia
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NephroNet, Inc. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NN-007
Record Dates: First submitted 2022-08-23; First posted 2022-09-10 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: Chronic outpatient hemodialysis patients have high rates of rapid changes in potassium and other electrolytes critical to the generation cardiac arrythmias. A growing body of data suggests that intra-dialytic K+ levels fall to level of 2.0 or lower and are a potential major contributor to the generation of atrial fibrillation, bradycardia, and other clinically significant arrhythmias. We propose that raising the dialysate bath to 3.0 K+ from current standard of care levels of 2.0 K+ will reduce levels of hypokalemia-induced arrhythmias. We further propose that the use of sodium zirconium cyclosilicate (Lokelma) will ensure that secondary hyperkalemia is controlled following the introduction of the 3.0 K+ dialysate bath.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rate Atrial fibrillation - 2.0K+ dialysate bath wo/ Lokelma to crossover (Other): Sequence A: standard 2.0 K+/2.5 Ca++ dialysate with no Lokelma supplementation for two (2) months, followed by a cross-over to experimental 3.0 K+/2.5 Ca++ dialysate with 5 grams powder oral suspension Lokelma supplementation (on off-dialysis days) for two (2) months.
  Each two-month treatment period (both 2.0 K+/2.5 Ca++ dialysate and 3.0 K+/2.5 Ca++ dialysate with Lokelma sequences) will be preceded by a two-week run-in period, to allow the patient to adapt to the new dialysate bath. While receiving the higher K+ dialysate, patient will be treated on off-dialysis days (4 days/week) with Lokelma, titrated to maintain K+ between 4.0 and 5.5 mEq/L. Refer to section 7.2 for the initial dose and frequency details.
  Interventions: Drug: LOKELMA 5 GM Powder for Oral Suspension
- Rate Atrial fibrillation - 3.0K+ dialysate bath w/ 5 grams Lokelma to crossover (Other): • Sequence B: experimental 3.0 K+/2.5 Ca++ dialysate with 5 grams Lokelma supplementation (on off-dialysis days) for two (2) months, followed by standard 2.0 K+/2.5 Ca++ dialysate with no Lokelma supplementation for two (2) months.
  Each two-month treatment period (both 2.0 K+/2.5 Ca++ dialysate and 3.0 K+/2.5 Ca++ dialysate with Lokelma sequences) will be preceded by a two-week run-in period, to allow the patient to adapt to the new dialysate bath. While receiving the higher K+ dialysate, patient will be treated on off-dialysis days (4 days/week) with Lokelma, titrated to maintain K+ between 4.0 and 5.5 mEq/L. Refer to section 7.2 for the initial dose and frequency details.
  Interventions: Drug: LOKELMA 5 GM Powder for Oral Suspension

INTERVENTIONS:
Drug: LOKELMA 5 GM Powder for Oral Suspension — Patients will use Lokelma supplementation on off-dialysis days (4 days/week) while receiving hemodialysis with 3.0 K+/2.5 Ca++ mEq dialysate bath. The individual starting dose will be 5.0 grams, and may be titrated weekly in 5.0 gram increments up to 15.0 grams to maintain K+ between 4.0 and 5.5 mEq/L.

SUMMARY:
A Prospective, RanDomized, Multi-Center, Open-Label, Cross-Over Study of Sodium Zirconium Cyclosilicate to Control Interdialytic HyperkalemiA Following Augmentation of Dialysate Potassium: Efficacy to Reduce the Incidence of Post-Dialysis Atrial Fibrillation and Clinically SignificanT Cardiac Arrhythmias - ADAPT Trial

DETAILED DESCRIPTION:
This is a prospective, open-labelled, randomized, 2x2 cross-over design study of 88 patients with end stage renal disease (ESRD) receiving routine out-patient dialysis using a standard 2.0 potassium ion (K+)/2.5 calcium ion (Ca++) dialysate bath. The overall aim of the study is to determine whether converting stable hemodialysis patients from a "standard" 2.0 K+/2.5 Ca+ dialysate (without Lokelma) to a 3.0 K+/2.5 Ca++ mEq dialysate supplemented with the orally administered potassium binder sodium zirconium cyclosilicate (Lokelma) to treat interdialytic hyperkalemia will reduce the incidence and duration of post-dialysis atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Female or male aged above 18 years
* Patients with ESRD receiving hemodialysis three times per week for a minimum of 3 months
* Patients must have two (2) pre-dialysis K+ measurements between 5.1 and 6.5 mEq/L by Piccolo POCT following the long dialytic "weekends" (i.e., on two consecutive Mondays for patients on a Monday-Wednesday-Friday dialysis schedule or on two consecutive Tuesdays for patients on a Tuesday-Thursday-Saturday dialysis schedule) during screening, before insertion of the cardiac loop recorder.
* Female participants must be 1 year post-menopausal, surgically sterile, or using one highly effective form of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly.) They should have been stable on their chosen method of birth control for a minimum of 1 month before entering the study and willing to remain on the birth control until 4 weeks after the last dose.

Exclusion Criteria:

-

Exclusion Criteria Related to the Underlying Condition:

* Patients with a QTc(f) > 550 msec and/or Congenital long QT syndrome
* Patients with a Haemoglobin < 9 g/dl.
* Patients with any medical condition, including active, clinically significant infection or liver disease, that in the opinion of the investigator or Sponsor may pose a safety risk to a subject in this study, which may confound safety or efficacy assessment and jeopardize the quality of the data, or may interfere with study participation.
* Patient receiving peritoneal or home hemodialysis
* Patient receiving hemodialysis via a tunneled inferior vena cava (IVC) catheter and known central stenosis of access extremity
* Patient receiving outpatient hemodialysis for < 3 months
* Patient receiving outpatient hemodialysis for prolonged Acute Kidney Injury (AKI) and considered by the site Principal Investigator (PI) likely to achieve renal recovery within 6 months Note: Patients receiving out-patient hemodialysis for AKI for longer than 6 months with no demonstrable renal clearance can be screened for study participation.
* Patient currently receiving a 1.0 K+, 3.0 K+ dialysate bath and unwilling to convert to a 2.0 K+/2.5 Ca++ dialysate bath
* Subject unwilling to convert from a 2.0 K+ dialysate bath to a 3.0 K+ dialysate bath
* Two or more pre-dialysis K+ of < 5.1 or > 6.5 mEq/L measured by Piccolo POCT after the long dialytic "weekends" during screening Note: If one of the two screening pre-dialysis K+ levels is between 4.6 to 5.0 mEq/L or 6.6 to 7.0 mEq/L, the patient can undergo an additional whole blood Piccolo POCT K+ measurement. Patients who fail the third whole blood Piccolo POCT K+ measurement will be considered ineligible for study participation. Note: Screen failures can be re-screened once to confirm eligibility in the study.
* Any documented whole blood Piccolo POCT K+ measurement that falls below 4.6 mEq/L or exceeds 7.0 mEq/l during the screening period
* Current use of a medication for treatment of hyperkalemia (e.g., Patiromer).
* Note: If a medication for treatment of hyperkalemia is stopped prior to or after the consenting process, the subject will undergo a one week washout prior to the first whole blood Piccolo POCT K+ measurement. Exclusion Criteria Related to Other Medical Conditions and Treatments:
* Anticipated life expectancy of 3 months duration
* Development of atrial fibrillation requiring hospitalization, medical therapy, anticoagulation, or cardioversion during study pre-screening or screening period
* Patient with a known placement of a dual or single chamber pacemaker
* Patient with an automatic implantable cardiac defibrillator (AICD)
* Patient with a LINQ implanted cardiac loop recorder with less than 6 months of battery life.
* Current use of amiodarone or other anti-arrhythmic therapy. Note: Patients on such medications must undergo a two week washout prior to the first whole blood Piccolo POCT K+ measurement.
* Known history of cardiac arrhythmias due to prolonged QT syndrome
* Subject unwilling to receive an implanted LINQ cardiac loop recorder (unless 6 months are remaining in their previously implanted device).
* Known active drug abuse
* Positive hepatitis C polymerase chain reaction (PCR) test with active viral deoxyribonucleic acid (DNA) shedding or chronic active hepatitis B as evidenced by detectable surface antigen from standard of care routine dialysis labs. Note: Patients with negative PCR DNA testing for either hepatitis B or C will be allowed to participate in the study.
* Known to have tested positive for human immunodeficiency virus (HIV) from standard of care routine dialysis labs.
* For women only: currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
* Patients with known and/or active severe constipation, bowel obstruction or impaction, including abnormal post-operative bowel motility disorders or diabetic gastroparesis Exclusion Criteria Related to the Investigational Product (IP):
* Known hypersensitivity to sodium zirconium cyclosilicate (Lokelmaâ).

Other/General Exclusion Criteria:

* Previous randomization in the present study. Note: Screen failures can be re-screened once to confirm eligibility in the study.
* Participation in another interventional (non-observational) clinical study within 4 weeks prior to enrollment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The change in atrial Fibrillation events | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To demonstrate whether increasing the K+ concentration in a standard hemodialysis bath from 2.0 K+ /2.5 Ca++ to a 3.0 K+ /2.5 Ca++ composition with SZC will reduce the incidence of atrial fibrillation events.

SECONDARY OUTCOMES:
Frequency and duration of CSCAs (bradycardia, ventricular tachycardia and/or asystole) | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To access whether the incidence and duration of post-dialysis CSCAs (defined as bradycardia, ventricular tachycardia and/or asystole) observed during experimental treatment will be reduced compared to standard treatment.
Whether or not K+ outside of the 4.0 to 5.5 mEq/L safety range (Yes/No binary outcome measure). | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To determine whether the addition of oral sodium zirconium cyclosilicate (Lokelmaâ) during the 2-month treatment phase with the 3.0 K+ /2.5 Ca++ dialysate bath will reduce risk of weeks outside the "K+ safety range" of 4.0 to 5.5 mEq/L compared to the 2-month treatment phase with the 2.0 K+ /2.5 Ca++ dialysate bath.

OTHER OUTCOMES:
Total number of hypokalemic events defined as Piccolo POCT or laboratory-measured K+ of < 3.5 mEq/L. | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To evaluate whether the use of oral sodium zirconium cyclosilicate (Lokelmaâ) during periods when patients are receiving a 3.0 K+ /2.5 Ca++ dialysate bath is associated with hypokalemic events defined as K+ <3.5 mEq/L.
Number of events (measured promptly prior to the termination of dialysis) where a Piccolo POCT measurement of K+ is < 3.5 mEq/L OR Ca++ is < 7.0 mEq/L, OR Mg++ is < 2.0 mg/dl, OR a PO4 level is <3.0 mEq/L | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To determine the levels of K+ , Mg++, calcium and PO4 during dialysis (measured promptly prior to the termination of dialysis) during experimental treatment compared to standard treatment.
Frequencies of AEs, SAEs, and withdrawals due to AEs, with focus on treatment-related events. | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To evaluate the safety and tolerability of the experimental treatment compared to standard treatment based on the frequency of reported adverse experiences.
Correlation between PBUTs (IS, PCS, and ADMA) and the frequency of atrial fibrillation events. | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To evaluate the relationship between proteinbound uremic toxins (PBUTs) and atrial fibrillation rates. PBUTs such indoxyl sulfate (IS) and p-Cresol. sulfate (PCS) can induce atrial fibrillation
Correlation between electrolyte levels and clinical events (intradialytic hypotension, muscle cramping, and cardiac events). Correlation between electrolytes falling below threshold levels | 8-week Treatment Phase-1 and the 8-week Treatment Phase-2 dialysate cross-over periods
  To determine whether the levels of K+, Mg++, calcium and PO4 (measured promptly prior to the termination of dialysis) correlate with the incidence of clinical events, including intradialytic hypotension, muscle cramping, and cardiac events (defined as atrial fibrillation, bradycardia, ventricular tachycardia, and asystole). We will also evaluate whether the 3.0 K+ dialysate reduces the rates of these clinical events.

CONTACTS AND LOCATIONS:
Overall Officials: James Tumlin, MD, Principal Investigator — NephroNet, Inc.; Jeremy Whitson, BS, Study Director — NephroNet, Inc.
Locations (5):
- United States (5):
  - Balboa Research, La Jolla, California
  - Georgia Nephrology DBA Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - Nephrology Associates of Northern Illinois and Indiana (NANI), Fort Wayne, Indiana
  - Clinical Research Consultants, Kansas City, Missouri
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT05535920/Prot_000.pdf